CLINICAL TRIAL: NCT02334306
Title: A Phase 2a, Randomized, Placebo Controlled, Proof of Mechanism Study to Evaluate the Safety and Efficacy of AMG 557/MEDI5872 in Subjects With Primary Sjögren's Syndrome
Brief Title: A Phase 2a, Randomized, Placebo Controlled, Study to Evaluate the Safety and Efficacy of AMG 557/MEDI5872 in Primary Sjögren's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5181C00001
Record Dates: First submitted 2014-12-12; First posted 2015-01-08 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-02

CONDITIONS: Primary Sjögren's Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MEDI5872 210 mg (Experimental): Participants will receive a fixed SC dose of 210 mg MEDI5872 every week (QW) from Days 1 to 15 and then every 2 weeks (Q2W) from Days 29 to 85 in double-blind period. In open-label period, participants will continue dosing of MEDI5872 210mg Q2W from Days 99 to 183 and will receive an additional dose of blinded placebo on Day 106.
  Interventions: Biological: AMG 557/MEDI5872
- Placebo/MEDI5872 210 mg (Placebo Comparator): Participants will receive a SC dose of placebo matching with MEDI5872 QW on Days 1, 8, and 15 and then Q2W from Days 29 to 85 in double-blind period. In open-label period, participants will receive a fixed SC dose of 210 mg MEDI5872 QW (Days 99 to 113) and Q2W (Days 127 to 183) in open-label period.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AMG 557/MEDI5872 — Participants will receive a fixed SC dose of 210 mg MEDI5872 (AMG 557/MEDI5872) QW for 3 weeks (Days 1 to 15) and then Q2W for 9 weeks (Days 29 to 85) in double-blind period of the study. In open-label period, all participants from double-blind period will receive a fixed SC dose of 210 mg MEDI5872 from Day 99 to Day 183 (QW from Days 99 to 113 for participants from Placebo arm and on Days 99 and 113 for participants from MEDI5872 210 mg arm; and Q2W from Days 127 to 183 for participants from both arms).
  Arms: MEDI5872 210 mg
Other: Placebo — The SC dose of placebo every week for 3 weeks (Days 1 to 15) and then every 2 weeks for 9 weeks (Days 29 to 85) in double-blind period of the study. In open-label period, an additional dose of blinded placebo will be administered on Day 106 for participants who will receive MEDI5872 210mg in double-blinded period.
  Arms: Placebo/MEDI5872 210 mg

SUMMARY:
A Phase 2a study to evaluate the efficacy and safety of AMG 557/MEDI5872 in Primary Sjögren's Syndrome

DETAILED DESCRIPTION:
This is a Phase 2a, multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the clinical and biologic efficacy, as well as the safety of SC doses of AMG 557/MEDI5872 in adult subjects with Primary Sjögren's Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 75 years at the time of signing the ICF.
* Fulfill American-European Consensus Group (AECG) criteria for pSS
* ESSDAI score ≥ 6.
* Positive anti-SS-A and/or anti-SS-B autoantibodies and at least IgG > 13 g/L or RF level > upper limit of normal (ULN) or positive test for cryoglobulins
* Willingness to undergo protocol-required minor salivary gland biopsies.
* Negative TB test during screening
* Immunization up to date as determined by local standard of care.

Exclusion Criteria:

* Previous treatment with AMG 557/MEDI5872.
* Evidence of signs or symptoms of a viral, bacterial, or fungal infection within 2 weeks (14 days) prior to randomization (Day 1) according to the assessment of the investigator; any infection requiring IV antibiotic or antiviral treatment within 8 weeks of randomization (Day 1); history of herpes zoster within 3 months prior to randomization (Day 1).
* Evidence of significant renal insufficiency
* Positive test at screening for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) antibody.
* Prior administration of any of the following:

  1. Belimumab in the past 6 months prior to randomization (Day 1);
  2. Rituximab in the past 12 months or CD19+ B cells < 5/µL if rituximab treatment was more than 12 months prior to randomization (Day 1);
  3. Abatacept in the past 6 months prior to randomization (Day 1);
  4. Tumor necrosis factor inhibitors (adalimumab, certolizumab, etanercept, golimumab, infliximab) in the past 3 months prior to randomization (Day 1);
  5. Tocilizumab in the past 3 months prior to randomization (Day 1);
  6. Cyclophosphamide (or any other alkylating agent) in the past 6 months prior to randomization (Day 1); cyclosporine (except for eye drops), tacrolimus, sirolimus, mycophenolate mofetil, azathioprine, or leflunomide in the past 3 months prior to randomization (Day 1).
* Receiving any of the following:

  1. Corticosteroids: > 10 mg/day oral prednisone (or equivalent); Any change or initiation of new dose within 4 weeks prior to signing the ICF through randomization (Day 1); Intramuscular, IV, or intra-articular corticosteroids within 4 weeks prior to signing the ICF through randomization (Day 1); Any change or initiation of new dose of topical corticosteroids within 2 weeks prior to signing the ICF through randomization (Day 1);
  2. Antimalarials: any increase or initiation of new dose of antimalarials (eg, chloroquine, hydroxychloroquine, quinacrine) within 12 weeks prior to signing the ICF through randomization (Day 1).
  3. Methotrexate: > 20 mg/week methotrexate; Any change or initiation of new dose of methotrexate within 4 weeks prior to signing the ICF through randomization (Day 1); Any change in route of administration.
  4. Any increase or initiation of new dose of regularly scheduled nonsteroidal anti inflammatory drugs (NSAIDs) within 2 weeks prior to signing the ICF through randomization (Day 1).
  5. Cevimeline or pilocarpine and cyclosporine eye drops (Restasis): any increase or initiation of new doses within 2 weeks prior to signing the ICF through randomization (Day 1).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-06-08 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Dall'Era, MD, Principal Investigator — University of California, San Francisco; Ghaith Noaiseh, MD, Principal Investigator — University of Pittsburgh
Locations (12):
- United States (3):
  - Research Site, San Francisco, California
  - Research Site, Bethesda, Maryland
  - Research Site, Pittsburgh, Pennsylvania
- France (5):
  - Research Site, Brest
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Lille
  - Research Site, Paris
  - Research Site, Strasbourg
- Research Site, Stockholm, Sweden
- United Kingdom (3):
  - Research Site, London
  - Research Site, Newcastle upon Tyne
  - Research Site, Swindon

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3677&filename=SAP%20D5181C00001%20amendment%201_redact.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3677&filename=SAP%20PDF-%20a.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3677&filename=protocol-d5181c00001-amendment-4-clean_CLM%20redact_Redacted%20PDFA.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted across 4 countries (France, United Kingdom, Sweden, and the United States).
Pre-assignment Details: A total of 59 participants were screened in the study. Of which, 27 participants were screen failures and 32 participants were randomized and enrolled in study. The results are posted per the data of primary efficacy analysis last participant last visit date.
Groups:
- Placebo/MEDI5872 210 mg: Participants received a subcutaneous (SC) dose of placebo matching with MEDI5872 every week (QW) for 3 weeks (Days 1, 8, and 15) and then every 2 weeks (Q2W) for next 9 weeks (Days 29 to 85) in double-blind period of the study. In open-label period, participants received MEDI5872 QW from Days 99 to 113 and Q2W from Days 127 to 183.
- MEDI5872 210 mg/MEDI5872 210 mg: Participants received a fixed SC dose of 210 mg MEDI5872 every week (QW) for 3 weeks (Days 1 to 15) and then every 2 weeks (Q2W) for next 9 weeks (Days 29 to 85) in double-blind period of the study. In open-label period, participants continued dosing of MEDI5872 210mg Q2W from Days 99 to 183 and received an additional dose of blinded placebo on Day 106.
Period: Double-blind Period
Arm/Group | Placebo/MEDI5872 210 mg | MEDI5872 210 mg/MEDI5872 210 mg
Started | 16 | 16
Completed | 15 | 14
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Open-label Period
Arm/Group | Placebo/MEDI5872 210 mg | MEDI5872 210 mg/MEDI5872 210 mg
Started | 15 | 14
Completed | 15 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/MEDI5872 210 mg | MEDI5872 210 mg/MEDI5872 210 mg | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The As-treated population included all treated participants, grouped according to actual treatment received.
  Years | 50.2 (12) | 51.1 (14.3) | 50.7 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 15 | 13 | 28
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in European League Against Rheumatism Sjogren's Syndrome Disease Activity Index (ESSDAI) Score at Day 99
Description: The European League Against Rheumatism Sjogren's Syndrome Disease Activity Index (ESSDAI) is a clinical index that measures Sjogren's syndrome disease activity. A physician scores the disease activity level of 12 organ-specific domains (constitutional, lymphadenopathy, articular, muscular, cutaneous, glandular, pulmonary, renal, peripheral nervous system, central nervous system, hematological, and biological). Each domain is assessed for activity level in 3 or 4 levels (i.e., no, low, moderate, high) according to their severity (no disease activity equals to 0 and for high disease activity the domain score equals 3 or 4). Each domain is assigned a weight between 1 and 6, and the domain score is multiplied by the domain weight. Overall score is calculated as sum of all individual weighted domain scores (ranges from 0 (best) to 123 (worst activity). A higher score indicates worsening of the disease. Adjusted mean change and standard error are presented.
Time Frame: Baseline (Day 1 predose) and Day 99
Population: Intent-to-treat (ITT) population included all randomized and treated participants, grouped according to assigned treatment. The "Overall Number of Participants Analyzed" denotes the number of participants evaluated for this outcome measure.
Measure: Mean (Standard Error); unit: Scores on a scale
Groups:
- Placebo: Participants received a subcutaneous (SC) dose of placebo matching with MEDI5872 every week (QW) for 3 weeks (Days 1, 8, and 15) and then every 2 weeks (Q2W) for next 9 weeks (Days 29 to 85) in double-blind period of the study.
- MEDI5872 210 mg: Participants received a fixed SC dose of 210 mg MEDI5872 every week (QW) for 3 weeks (Days 1 to 15) and then every 2 weeks (Q2W) for next 9 weeks (Days 29 to 85) in double-blind period of the study.
Arm/Group | Placebo | MEDI5872 210 mg
Number analyzed (Participants) | 16 | 13
Scores on a scale | -2.3 (0.8) | -3.8 (0.9)
Statistical Analysis 1: Comparison: Placebo vs MEDI5872 210 mg; Test type: Superiority; p = 0.262, ANCOVA; Mean Difference (Net) = -1.4, 90% CI 2-sided [-3.6 to 0.7], Standard Error of Mean 1.3 — Adjusted mean difference for MEDI5872 210 mg:Placebo was calculated with associated 90% confidence interval and p-value

2. Secondary Outcome: Ratio to Baseline in Peripheral Blood Biomarkers at Day 99
Description: The peripheral blood biomarkers included total plasma cell levels (including plasma blast levels) and T follicular helper (TFH) cells. Adjusted geometric mean ratio to baseline and standard error (log) are presented.
Time Frame: Baseline (Day 1 predose) and Day 99
Population: The ITT population included all randomized and treated participants, grouped according to assigned treatment.
Measure: Geometric Mean (Standard Error); unit: Ratio
Arm/Group | Placebo | MEDI5872 210 mg
Number analyzed (Participants) | 16 | 16
Ratio
  Plasma Cell Levels | 0.70 (0.24) | 0.65 (0.24)
  TFH Cells | 0.94 (0.27) | 0.62 (0.27)
Statistical Analysis 1: Comparison: Placebo vs MEDI5872 210 mg; For plasma cell levels; Test type: Superiority; p = 0.820, ANCOVA; Mean Difference (Net) = 0.93, 90% CI 2-sided [0.52 to 1.64], Standard Error of Mean 0.33 — Adjusted Geometric mean ratio for MEDI5872 210 mg:Placebo was calculated with associated 90% confidence interval, SE (log), and p-value
Statistical Analysis 2: Comparison: Placebo vs MEDI5872 210 mg; For TFH cells; Test type: Superiority; p = 0.291, ANCOVA; Median Difference (Net) = 0.65, 90% CI 2-sided [0.33 to 1.28], Standard Error of Mean 0.40 — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Ratio to Baseline in Minor Salivary Gland Tissue Biomarkers at Day 99
Description: The minor salivary gland biopsy biomarkers included total plasma cell levels, CD4/ inducible T-cell costimulator (ICOS) TFH cells, and PD-1/ICOS TFH cells. Adjusted geometric mean ratio to baseline and standard error (log) are presented.
Time Frame: Baseline (Day 1 predose) and Day 99
Population: The ITT population included all randomized and treated participants, grouped according to assigned treatment.
Measure: Geometric Mean (Standard Error); unit: Ratio
Arm/Group | Placebo | MEDI5872 210 mg
Number analyzed (Participants) | 16 | 16
Ratio
  Total Plasma Cells: number analyzed (Participants) | 9 | 11
  Total Plasma Cells | 1.32 (0.13) | 1.15 (0.11)
  CD4/ICOS TFH Cells: number analyzed (Participants) | 9 | 11
  CD4/ICOS TFH Cells | 1.76 (0.21) | 0.75 (0.18)
  PD-1/ICOS TFH Cells: number analyzed (Participants) | 9 | 11
  PD-1/ICOS TFH Cells | 1.06 (0.19) | 1.07 (0.16)
Statistical Analysis 1: Comparison: Placebo vs MEDI5872 210 mg; For total plasma cells; Test type: Superiority; p = 0.440, ANCOVA; Mean Difference (Net) = 0.87, 90% CI 2-sided [0.65 to 1.18], Standard Error of Mean 0.17 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs MEDI5872 210 mg; For CD4/ICOS TFH cells; Test type: Superiority; p = 0.008, ANCOVA; Median Difference (Net) = 0.43, 90% CI 2-sided [0.26 to 0.70], Standard Error of Mean 0.28 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs MEDI5872 210 mg; For PD-1/ICOS TFH cells; Test type: Superiority; p = 0.972, ANCOVA; Median Difference (Net) = 1.01, 90% CI 2-sided [0.64 to 1.59], Standard Error of Mean 0.26 — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Ratio to Baseline in Focus Score at Day 99
Description: The focus score is a semi-quantitative assessment of focal lymphocytic sialoadenitis, which is defined as the presence of >= 1 dense aggregate of 50 or more lymphocytes in a 4 mm2 area. Higher numbers are associated with more inflammation.
Time Frame: Baseline (Day 1 predose) and Day 99
Population: The ITT population included all randomized and treated participants, grouped according to assigned treatment. The "Overall Number of Participants Analyzed" denotes the number of participants evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | MEDI5872 210 mg
Number analyzed (Participants) | 6 | 10
Ratio | 0.79 (0.53) | 0.96 (0.50)

5. Secondary Outcome: Change From Baseline in European League Against Rheumatism Sjogren's Syndrome Patient Reported Index (ESSPRI) Score at Day 99
Description: The European League Against Rheumatism Sjogren's Syndrome Patient Reported Index (ESSPRI) is a patient-reported, subjective symptom index for primary Sjögren's syndrome. It consists of three questions covering the cardinal symptoms of Sjögren's syndrome: dryness, fatigue and pain (articular and/or muscular). Each domain scored on scale of 0-10 (0 =no symptom at all and 10 = worst symptom imaginable), and an overall score is calculated as the mean of the three individual domains where all domains carry the same weight. Adjusted mean change and standard error are presented.
Time Frame: Baseline (Day 1 predose) and Day 99
Population: The ITT population included all randomized and treated participants, grouped according to assigned treatment.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | MEDI5872 210 mg
Number analyzed (Participants) | 16 | 16
Scores on a scale | -1.0 (0.5) | -0.6 (0.5)
Statistical Analysis 1: Comparison: Placebo vs MEDI5872 210 mg; Test type: Superiority; p = 0.574, ANCOVA; Mean Difference (Net) = 0.4, 90% CI 2-sided [-0.8 to 1.6], Standard Error of Mean 0.7 — Adjusted mean difference for MEDI5872 210 mg:Placebo was calculated with associated 90% confidence interval and p-value

6. Secondary Outcome: Percentage of ESSDAI Responders at Day 99
Description: The ESSDAI is a clinical index that measures Sjogren's syndrome disease activity. A physician scores the disease activity level of 12 organ-specific domains (constitutional, lymphadenopathy, articular, muscular, cutaneous, glandular, pulmonary, renal, peripheral nervous system, central nervous system, hematological, and biological). Each domain is assessed for activity level in 3 or 4 levels (no, low, moderate, high) according to their severity (0=no disease activity and ¾ = high disease activity of the domain). Each domain is assigned a weight between 1 and 6, and the domain score is multiplied by the domain weight. Overall score is calculated as sum of all individual weighted domain scores (ranges from 0 [best] to 123 [worst activity]). Participants are considered to be an ESSDAI[x] responder as they achieved a reduction of x points or more in ESSDAI score, did not prematurely discontinue the study drug, and did not receive prohibited concomitant medications.
Time Frame: Baseline (Day 1 predose) and Day 99
Population: The ITT population included all randomized and treated participants, grouped according to assigned treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | MEDI5872 210 mg
Number analyzed (Participants) | 16 | 16
Percentage of participants
  ESSDAI [3] | 18.8 | 43.8
  ESSDAI [4] | 18.8 | 43.8
Statistical Analysis 1: Comparison: Placebo vs MEDI5872 210 mg; ESSDAI [3]; Test type: Superiority; p = 0.252, Fisher Exact; Difference in percentages = 25, 90% CI 2-sided [-3.1 to 50.9]
Statistical Analysis 2: Comparison: Placebo vs MEDI5872 210 mg; ESSDAI[4]; Test type: Superiority; p = 0.252, Fisher Exact; Difference in precentages = 25, 90% CI 2-sided [-3.1 to 50.9]

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs were collected from Day 1 (postdose) until Day 99 for 'Placebo' arm and Day 296 for 'Any MEDI5872 210 mg' arm that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Placebo arm: Day 1 (postdose) through Day 99 (predose); Any MEDI5872 210 mg arm: Day 1 (postdose) through Day 296 for MEDI5872 210 mg arm, and Day 99 (postdose) through Day 296 for participants who received placebo at double-blind period
Population: Placebo: As-treated population (participants grouped per actual treatment received).
  Any MEDI5872 210 mg: Any MEDI5872 population (participants received at least 1 dose of MEDI5872 either in double-blind and/or open-label). 1 participant from 'Placebo' discontinued treatment before Day 99 and didn't receive MEDI5872 dose in open-label period.
Measure: Count of Participants; unit: Participants
Groups:
- Any MEDI5872 210 mg: Participants received at least one dose of MEDI5872 treatment either during double-blind and/or open-label period of the study.
  In double-bind period, participants received a fixed SC dose of 210 mg MEDI5872 QW for 3 weeks (Days 1, 8, and 15) and then every Q2W for 9 weeks (Days 29 to 85).
  In open-label period, participants who received MEDI5872 210mg in double-blinded period received MEDI5872 210mg on Days 99 and Day 113; and participants who received placebo in double-blinded period received MEDI5872 210mg QW from Days 99 to 113, later all participants received MEDI5872 210mg Q2W from Days 127 to 183 and were followed up till Day 296.
Arm/Group | Placebo | Any MEDI5872 210 mg
Number analyzed (Participants) | 16 | 31
Participants
  Any TEAEs | 14 | 29
  Any TESAEs | 0 | 1

8. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: An AESI (serious or non-serious) was one of scientific and medical interest specific to understanding of study drug and may have required close monitoring and rapid communication by investigator to the sponsor. The AESIs for this study were hepatic function abnormality meeting the definition of Hy's law, new or reactivated tuberculosis infection, malignancy, and hypersensitivity and anaphylactic reactions. Treatment-emergent AESIs were collected from Day 1 (postdose) until Day 99 for 'Placebo' arm and Day 296 for 'Any MEDI5872 210 mg' arm.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Any MEDI5872 210 mg
Number analyzed (Participants) | 16 | 31
Participants | 1 | 6

ADVERSE EVENTS:
Time Frame: Placebo arm: Day 1 (postdose) through Day 99 (predose); Any MEDI5872 210 mg arm: Day 1 (postdose) through Day 296 for MEDI5872 210 mg arm, and Day 99 (postdose) through Day 296 for participants who received placebo at double-blind period 1 participant from 'Placebo' arm discontinued treatment before Day 99, didn't receive MEDI5872 dose and entered in safety follow-up period.
Arm/Group | Placebo | Any MEDI5872 210 mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/31
Other Adverse Events (participants affected / at risk) | 14/16 | 29/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Any MEDI5872 210 mg (N=31)
Small intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Any MEDI5872 210 mg (N=31)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 2 (4)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (5)
Dental caries (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip blister (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Parotid gland enlargement (Gastrointestinal disorders) | 1 (2) | 1 (1)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue blistering (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (3)
Fatigue (General disorders) | 0 (0) | 2 (2)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 2 (2) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 2 (7)
Injection site haematoma (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 3 (5)
Injection site rash (General disorders) | 0 (0) | 4 (5)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Local swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Vaccination site reaction (General disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 2 (2)
Genital candidiasis (Infections and infestations) | 0 (0) | 1 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 3 (7)
Paronychia (Infections and infestations) | 0 (0) | 2 (2)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Serratia infection (Infections and infestations) | 0 (0) | 1 (1)
Tongue fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 8 (8)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (6)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (3) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)
Accidental device ingestion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Tooth avulsion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 1 (1)
Calcium deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 5 (8)
Paraesthesia (Nervous system disorders) | 1 (2) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Stress (Psychiatric disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (4)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (7)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 0 (0) | 2 (4)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT02334306/SAP_000.pdf
  • Study Protocol (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT02334306/Prot_001.pdf